CLINICAL TRIAL: NCT00292721
Title: Effects of Celecoxib on Restenosis After Percutaneous Coronary Intervention and Evolution of Atherosclerosis (COREA) Trial
Brief Title: Effects of Celecoxib After Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul national university hostpial, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 134-가-37
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Celecoxib (Active Comparator)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — celecoxib: loading and maintenance for 6 months
  Arms: Celecoxib

SUMMARY:
Several studies including ours have reported that celecoxib improves endothelium-dependent vasodilation and reduces inflammation and neointimal hyperplasia. Our hypothesis is that celecoxib may reduce the late luminal loss after coronary stent implantation (paclitaxel-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease with at least 1 de novo lesion greater than 50% stenosis on coronary angiography

Exclusion Criteria:

* Acute ST elevation MI
* Left main disease
* Contraindications to aspirin, clopidogrel or celecoxib
* Severe congestive heart failure
* Expected survival < 2 years
* Hepatic dysfunction
* Currently taking NSAIDs or any COX-2 inhibitor
* Renal dysfunction
* Use of warfarin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2004-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Late luminal loss at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Chung JW, Yang HM, Park KW, Lee HY, Park JS, Kang HJ, Cho YS, Youn TJ, Koo BK, Chae IH, Choi DJ, Oh BH, Park YB, Kim HS. Long-term outcome of adjunctive celecoxib treatment after paclitaxel-eluting stent implantation for the complex coronary lesions: two-year clinical follow-up of COREA-TAXUS trial. Circ Cardiovasc Interv. 2010 Jun 1;3(3):243-8. doi: 10.1161/CIRCINTERVENTIONS.109.889881. Epub 2010 May 18. PMID 20484099
- [Derived] Koo BK, Kim YS, Park KW, Yang HM, Kwon DA, Chung JW, Hahn JY, Lee HY, Park JS, Kang HJ, Cho YS, Youn TJ, Chung WY, Chae IH, Choi DJ, Oh BH, Park YB, Kim HS. Effect of celecoxib on restenosis after coronary angioplasty with a Taxus stent (COREA-TAXUS trial): an open-label randomised controlled study. Lancet. 2007 Aug 18;370(9587):567-74. doi: 10.1016/S0140-6736(07)61295-1. PMID 17707751